CLINICAL TRIAL: NCT02317978
Title: Evaluation of the Role of Follicular Sensitivity Index in the Prediction of IVF/ICSI Outcome
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer of Gynecology and Obstetrics, Cairo University
Other Study IDs: Sub8
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Subfertility
MeSH Terms: conditions — Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Subfertility without polycystic ovarian syndrome: The records of all women with infertility who had IVF/ICSI without polycystic ovarian syndrome (PCO) will be reviewed
  Interventions: Procedure: ICSI

INTERVENTIONS:
Procedure: ICSI — records of women who had ICSI will be reviewed and analysed for determining FSI

SUMMARY:
Records of women who had in vitro fertilization (IVF) or intra-cytoplasmic sperm injection (ICSI) in Dar AlTeb sub-fertility center will be reviewed and the follicular sensitivity index (FSI) will be calculated and correlated with pregnancy.

DETAILED DESCRIPTION:
The investigators study is a retrospective cohort study. Records of women who had in vitro fertilization (IVF) or intra-cytoplasmic sperm injection (ICSI) in Dar AlTeb sub-fertility center from January 2010 to December 2013 will be reviewed. All records with missing data will be excluded.

Triptorelin 0.1mg (Decapeptyl® Ferring, Germany) was used for pituitary down-regulation. It was given 7 days after the expected time of ovulation in women with regular cycles. Women with irregular cycles were given combined oral contraceptive pills and triptorelin was started on day 21 after starting the pills. On the second day of menstruation serum FSH, LH, Prolactin and Oestradiol were assessed and the antral follicular count (AFC) was assessed using a vaginal ultrasound scan. AFC will be defined as the number of follicles measuring 3-10mm.

Controlled ovarian hyperstimulation (COH) was started on the 2nd day of menstruation using human menopausal gonadotrophin (HMG) (Merional® IBSA, Switzerland). The initial dose ranged between 150-300 IU/day. The COH drug dose was adjusted according to the patient's response guided by number and size of the follicles in addition to serum E2 values. COH was continued until at least 3 follicles ≥17mm were obtained. This was followed by the administration of Human chorionic gonadotrophin (HCG) (Choriomon®, IBSA, Switzerland) 10000 IU. On the day of HCG administration, ovarian ultrasound scan will be performed using a transvaginal probe and the Preovulatory follicle count (PFC) was assessed, (PFC) was defined as number of follicles measuring≥16mm. FSI will be calculated as (FSI =PFC*10000/AFC*Total dose of FSH) Oocyte retrieval was guided by transvaginal ultrasound and was done 34-36 hours following HCG administration. Fertilization was done by ICSI. 16-18 hours later, fertilization was confirmed by the presence of 2 pronuclei.

The procedure was cancelled if less than 3 follicles ≥17 mm in size are present 12 days after starting FSH despite doses reaching 450 IU. The cycle was also cancelled if there is risk of ovarian hyperstimulation like massive ovarian enlargement or serum estradiol exceeds 3000pg/L The quality of embryos was assessed at day 3 according to the number and evenness of blastomeres in addition to the percentage of fragmentation. Embryos were classified into 3 groups: Excellent embryos containing 6-8 even blastomeres with <10% fragmentation, moderate embryos containing 6-8 even or uneven blastomeres with 10-20% fragmentation, and poor quality embryos containing less than 6 blastomeres or >20% fragmentation.

Embryo transfer was done on the 5th day after oocyte retrieval for couples who had IVF/ICSI. If possible, 2 embryos were transferred and cryopreservation of the remaining embryos was offered.

Luteal support was given in the form of progesterone vaginal tablets (Prontogest® IBSA, Switzerland) 400mg/day starting from the day of oocyte retrieval. A pregnancy test was done 2 weeks after embryo transfer and clinical pregnancy was defined as the presence of an intrauterine gestational sac 5 weeks after embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* IVF/ICSI

Exclusion Criteria:

* Missing data
* Cancelled cycles.
* Polycystic ovarian syndrome.

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The records of women who had IVF/ICSI without PCO will be reviewed to calculate the FSI.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy | 5 weeks after embryo transfer
  FSI values will be classified into 3 groups: High, moderate and low. The proportion of women achieving a clinical pregnancy will be compared among the 3 groups. clinical pregnancy will be defined as the presence of an intrauterine gestational sac 5 weeks after embryo transfer.

SECONDARY OUTCOMES:
Number of retrieved oocytes | one hour after ovum pick-up
  FSI values will be classified into 3 groups: High, moderate and low. the number of retrieved oocytes will be compared among the groups

CONTACTS AND LOCATIONS:
Locations (1):
- Dar AlTeb subfertility centre, Cairo, Egypt

REFERENCES:
- [Background] Zhang N, Hao CF, Zhuang LL, Liu XY, Gu HF, Liu S, Chen ZJ. Prediction of IVF/ICSI outcome based on the follicular output rate. Reprod Biomed Online. 2013 Aug;27(2):147-53. doi: 10.1016/j.rbmo.2013.04.012. Epub 2013 May 4. PMID 23768619
- [Background] Broer SL, Mol BW, Hendriks D, Broekmans FJ. The role of antimullerian hormone in prediction of outcome after IVF: comparison with the antral follicle count. Fertil Steril. 2009 Mar;91(3):705-14. doi: 10.1016/j.fertnstert.2007.12.013. Epub 2008 Mar 5. PMID 18321493
- [Background] Melo MA, Garrido N, Alvarez C, Bellver J, Meseguer M, Pellicer A, Remohi J. Antral follicle count (AFC) can be used in the prediction of ovarian response but cannot predict the oocyte/embryo quality or the in vitro fertilization outcome in an egg donation program. Fertil Steril. 2009 Jan;91(1):148-56. doi: 10.1016/j.fertnstert.2007.11.042. Epub 2008 May 2. PMID 18455166